CLINICAL TRIAL: NCT06677762
Title: A Retrospective Study on the Efficacy of Irreversible Electroporation Ablation Combined With Anti-PD(L)1 Therapy for Locally Advanced Pancreatic Cancer
Brief Title: Irreversible Electroporation Ablation Combined With Anti-PD(L)1 Therapy for Locally Advanced Pancreatic Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-421
Record Dates: First submitted 2024-10-30; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; irreversible electroporation; PD-(L)1
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Preserve the tissue and paraffin from pancreatic cancer and liver metastasis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IRE group: Patients who receive IRE ablation only
  Interventions: Procedure: Irreversible electroporation
- IRE+anti-PD（L）1: Patients who receive IRE ablation combined with anti-PD（L）1
  Interventions: Procedure: Irreversible electroporation

INTERVENTIONS:
Procedure: Irreversible electroporation — Irreversible electroporation ablation is an interventional ablation method, while anti-PD(L)1 is an immunotherapy.

SUMMARY:
Pancreatic cancer is a highly lethal malignant tumor of the digestive tract, especially local advanced pancreatic cancer (LAPC), which often loses the opportunity for surgical resection at the time of diagnosis. LAPC patients are often accompanied by tumor invasion of key anatomical structures such as major blood vessels, and traditional treatment methods such as radiotherapy and chemotherapy can slow down the progression of the disease, but the effect is limited, and the overall survival rate is still very low. There is a lack of effective treatment options for LAPC, especially in local control and prolonging survival, which exists a major limitation.

The surgical resection rate is low in LAPC, and the postoperative recurrence rate is high, and traditional radiotherapy and chemotherapy are difficult to completely eliminate the tumor. Immunotherapy has achieved breakthroughs in other tumors such as melanoma and non-small cell lung cancer, but the effect is limited in pancreatic cancer due to the immunosuppressive state of the tumor microenvironment (TME), which limits the efficacy of immunotherapy. In addition, the high invasiveness and rapid progression of pancreatic cancer further aggravates the treatment challenge.

Recent studies have shown that local ablation techniques such as irreversible electroporation (IRE) ablation not only can effectively ablate local tumors, but also may destroy the structural integrity of tumor cells, release tumor-associated antigens, and enhance the anti-tumor effect of the immune system. Therefore, IRE ablation may provide local control of pancreatic cancer for patients. At the same time, the combination of immune checkpoint inhibitors such as anti-PD(L)1 inhibitors may enhance the immune response in the tumor microenvironment and further improve the therapeutic effect. This combined treatment regimen is expected to overcome the limitations of single therapy and provide a new treatment strategy for local advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* The pathological diagnosis is local advanced pancreatic cancer that cannot be removed by surgery;
* Received IRE ablation treatment alone or in combination with anti-PD-1 or anti-PD-L1 immune inhibitors;
* Aged 18 years or older, gender is not limited, ECOG score 0-2;
* Have complete medical records and imaging follow-up records;
* At least 6 months of follow-up data.

Exclusion Criteria:

* Patients with other malignant tumors or severe immune system disorders;
* Patients who cannot complete follow-up or have missing data;
* Patients who have previously received immunotherapy without effect;
* Patients with severe organ dysfunction or who cannot tolerate further - - treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Include patients with locally advanced pancreatic cancer who received IRE ablation and combined anti-PD(L)1 treatment at Ruijin Hospital from January 2017 to December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
OS，Overall Survival | From the time of treatment to the death from any cause, assessed up to 35 months
  The patient received treatment until death.
PFS，Progress Free Survival | From the time of treatment to tumor progression or date of death from any cause, whichever came first, assessed up to 35 months
  Time of progression or death of the patient

SECONDARY OUTCOMES:
ORR，Objective response rate | From the time of treatment to tumor response or date of death from any cause, whichevercame first, assessed up to 35 months
  The proportion of patients whose tumor size decreases to a predetermined value and can maintain that minimum value for the required duration.

IPD SHARING:
Plan to Share IPD: No